CLINICAL TRIAL: NCT00831428
Title: A Pilot Study to Identify the Prevalence of Exercise- Induced Asthma and Rhinitis in Scottish Swimmers, Using Mannitol Challenge as a Screening Tool.
Brief Title: Screening Scottish Swimmers for Asthma and Rhinitis
Acronym: CLE004
Status: Completed | Type: Observational
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Other Study IDs: CLE004
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2011-09-23 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Asthma; Rhinitis
Keywords: asthma; rhinitis; swimmers; mannitol
MeSH Terms: conditions — Asthma; Rhinitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scottish swimming team
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is a screening study, not an interventional study

SUMMARY:
The Scottish National and District swimming teams will be screened for asthma and rhinitis using both mannitol challenge and sport-based exercise challenge.

ELIGIBILITY:
Inclusion Criteria:

* member of the Scottish national and district swimming team
* informed consent obtained

Exclusion Criteria:

* pregnant, lactating or planning to become pregnant
* concomitant use of medicines (prescribed, over-the-counter or herbal) that may interfere with the trial.
* any clinically significant medical condition, as deemed by the clinical investigators, which may endanger the health of the participant or jeopardise the protocol.
* inability to comply with the protocol.

Ages: 11 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Scottish national and district swimming teams
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karine L Clearie, MBBS, MRCP, Principal Investigator — Asthma and Allergy Research Group; Brian J Lipworth, MBchB, Study Director — Asthma and Allergy Research Group
Locations (1):
- The national swimming academy in Stirling, Stirling, Stirlingshire, United Kingdom

REFERENCES:
- [Result] Clearie KL, Williamson PA, Vaidyanathan S, Short P, Goudie A, Burns P, Hopkinson P, Meldrum K, Howaniec L, Lipworth BJ. Disconnect between standardized field-based testing and mannitol challenge in Scottish elite swimmers. Clin Exp Allergy. 2010 May;40(5):731-7. doi: 10.1111/j.1365-2222.2010.03461.x. Epub 2010 Mar 1. PMID 20214665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The scottish national and district teams were assessed during training weekends.
Pre-assignment Details: All members of the squad were offered the opportunity to take part.
Period: Overall Study
Arm/Group | Scottish Swimming Team
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Scottish Swimming Team
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 97
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 45
Region of Enrollment [Number; unit: participants]
  United Kingdom | 97

OUTCOME MEASURES:

1. Secondary Outcome: Mannitol Challenge
Time Frame: This test will be performed once on a district and once on a national squad training day
Reporting Status: Not Posted

2. Secondary Outcome: Sport-based Challenge
Time Frame: This test will be performed once on a district and once on a national squad training day
Reporting Status: Not Posted

3. Primary Outcome: Tidal Nitric Oxide
Time Frame: This test will be performed prior to entering the pool, and on exiting the pool
Population: Data from all participants was analysed
Measure: Geometric Mean (95% Confidence Interval); unit: ppb
Arm/Group | Scottish Swimming Team
Number analyzed (Participants) | 97
ppb | 18.7 [15.9 to 22.0]

4. Secondary Outcome: Nasal Nitric Oxide
Time Frame: This test will be performed prior to entering the pool, and on exiting the pool
Reporting Status: Not Posted

5. Secondary Outcome: Skin Prick Test
Time Frame: This test will be performed once on a district and once on a national squad training day
Reporting Status: Not Posted

6. Secondary Outcome: Mini Nasal Lavage
Time Frame: This test will be performed prior to entering the pool, and on exiting the pool
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Scottish Swimming Team
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes